CLINICAL TRIAL: NCT02567747
Title: Impact of Vaccination Against Pneumococcal Disease on the Morbidity of Acute Otitis Media in Colombian Children < 5 Years of Age
Brief Title: Vaccination Impact Against Pneumococcal Disease on Acute Otitis Media Morbidity in Colombian Children < 5 Years of Age
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 203127
Record Dates: First submitted 2015-09-28; First posted 2015-10-05 (Estimated); Last update posted 2019-06-10 (Actual); Status verified 2019-06

CONDITIONS: Acute Otitis Media; Pneumonia
Keywords: Colombia; otitis; Database; pneumonia
MeSH Terms: conditions — Otitis Media; Pneumonia; Otitis | interventions — Data Collection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Study cohort: The Total population will include all subjects included in the study. Only aggregated information will be collected for these subjects.
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — Data will be collected retrospectively for cases identified through RIPS*/ DANE** from 2008 until 2014 and through PAI*** from 2009 until 2014. *Registro Individual de Prestación de Servicios de Salud (RIPS) database (Health Service Provider Individual Registration Database), Columbia. **Departamento Administrativo Nacional de Estadística (DANE) database (The National Administrative Department of Statistics database), Columbia. ***Programa Ampliado de Immunizaciones (PAI) database (National Immunization Program database), Columbia.

SUMMARY:
The purpose of this study is to provide data on trends of morbidity due to Acute Otitis Media (AOM) (primary analysis) and morbidity and mortality due to pneumonia, and AOM related health care resources before and after the introduction of vaccination against pneumococcal disease within the Universal Mass Vaccination (UMV) in Colombia.

ELIGIBILITY:
Inclusion Criteria:

* Children aged less than five years with record of acute otitis media (with ICD-10 codes: H65 to H66) AND/OR.
* Children aged less than five years with record of pneumonia (with ICD-10 codes: J13 to J18) AND/OR.
* Children aged less than five years with any ICD-10 codes for respiratory diseases (J00-J99).

Exclusion Criteria:

• Not applicable

Max Age: 59 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: All eligible subjects (aggregated) captured by the selected national databases in Columbia.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2018-02-23 (Actual)

PRIMARY OUTCOMES:
Occurrence of reported cases of AOM in children below 5 years of age, in post-vaccination period compared to pre-vaccination period of PCV vaccination in UMV | Up to 7 years : from January 2008 to December 2014

SECONDARY OUTCOMES:
Occurrence of reported cases of AOM in children by morbidity, age group, and department in children in post-vaccination period compared to pre-vaccination period of PCV vaccination | Up to 7 years : from January 2008 to December 2014
  Morbidity including hospitalization, outpatient visits and ICD-10 code type, age groups including 0-24 months and 25-59 months strata.
Occurrence of reported cases of pneumonia and acute respiratory infections, overall and by morbidity, age groups, and department in children below 5 years of age before and after implementation of PCV vaccination into the UMV | Up to 7 years : from January 2008 to December 2014
  morbidity including hospitalization, outpatient visits and ICD-10 code type, age groups including 0-24 months and 25-59 months strata
Occurrence of reported deaths due to pneumonia and acute respiratory infections by age group (0-24 months and 25-59 months), department and overall in children below 5 years of age before and after implementation of PCV vaccination into the UMV | Up to 7 years : from January 2008 to December 2014
Occurrence of AOM related health care resources used and costs* before and after implementation of PCV vaccination into UMV by age group (0-24 months and 25-59 months) and overall | Up to 7 years : from January 2008 to December 2014
  * Cost calculation (e.g. medical procedures** , physician visits [outpatient/inpatient and length of stay]) will be extracted from Medical Procedure Cost Manual from the MOH for this analysis: http://www.fasecolda.com/index.php/ramos/soat/tarifas-y-coberturas/manual-tarifario-de-salud/. ** Tympanostomies/myringotomies, myringotomies with insertion of ventilation tubes, etc.
Total number of doses (complete or partial) of PCV vaccination administered in infants <1year of age after its introduction into the UMV program in Colombia. | Up to 7 years : from January 2008 to December 2014

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Bogotá, Colombia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Carrasquilla G, Porras-Ramirez A, Martinez S, DeAntonio R, Devadiga R, Talarico C, Caceres DC, Castrejon MM, Juliao P. Trends in all-cause pneumonia and otitis media in children aged <2 years following pneumococcal conjugate vaccine introduction in Colombia. Hum Vaccin Immunother. 2021 Apr 3;17(4):1173-1180. doi: 10.1080/21645515.2020.1805990. Epub 2020 Sep 23. PMID 32966144
- See also: Results for study 203127 can be found on the GSK Clinical Study Register — https://www.gsk-studyregister.com/study/5585